CLINICAL TRIAL: NCT03844776
Title: A Comparison of Single Preoperative Dose of Co-amoxiclav Versus Postoperative Full Course of Amoxicillin/ Co-amoxiclav in Prevention of Postoperative Complications in Dentoalveolar Surgery: a Randomized Controlled Trial
Brief Title: Preoperative Dose of Co-amoxiclav for Prevention of Postoperative Complications in Dentoalveolar Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taibah University (Other)
Responsible Party: Principal Investigator, Giath Gazal, Associate Professor, Taibah University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: IORG0008371
Record Dates: First submitted 2019-02-11; First posted 2019-02-18 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Infection
Keywords: dry socket; bleeding; swelling
MeSH Terms: conditions — Infections; Dry Socket; Hemorrhage | interventions — Amoxicillin-Potassium Clavulanate Combination; Acetaminophen; Saline Solution; Amoxicillin; Metronidazole

STUDY DESIGN:
Intervention Model Description: * Treatment 1: 0.9% normal saline irrigation immediately after the surgery with course of Amoxicillin 500 mg following the surgery for 5 days (control group)
  * Treatment 2: 625 mg Co-Amoxiclav and 1g paracetamol preoperatively and 0.2% chlorhexidine mouthwash immediately before the surgery but there is no additional course of antibiotic following the surgery.
  * Treatment 3: 0.9% normal saline irrigation immediately after the surgery with course of antibiotic Co-Amoxiclav for five days postoperatively
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Co-Amoxiclav postoperatively alone (Active Comparator): • Treatment 1: 0.9% normal saline irrigation immediately after the surgery with course of Co-Amoxiclav 625 mg 0.2% chlorhexidine mouthwash following the surgery for 5 days (control group)
  Interventions: Drug: Co-Amoxiclav; Drug: Chlorhexidine mouthwash; Drug: Normal saline
- Co-Amoxiclav preoperatively with Metronidazole postoperatively (Active Comparator): • Treatment 2: 625 mg Co-Amoxiclav and 1g Paracetamol preoperatively and 0.2% chlorhexidine mouthwash immediately before the surgery with course of Metronidazole 500 mg and 0.2% chlorhexidine mouthwash following the surgery for 5 days
  Interventions: Drug: Co-Amoxiclav; Drug: Paracetamol; Drug: Chlorhexidine mouthwash; Drug: Normal saline; Drug: Metronidazole
- Co-Amoxiclav preoperatively with amoxicillin postoperatively (Active Comparator): • Treatment 3: 625 mg Co-Amoxiclav and 1g Paracetamol preoperatively and 0.2% chlorhexidine mouthwash immediately before the surgery with course of amoxicillin 500 mg and 0.2% chlorhexidine mouthwash following the surgery for 5 days
  Interventions: Drug: Co-Amoxiclav; Drug: Paracetamol; Drug: Chlorhexidine mouthwash; Drug: Normal saline; Drug: Amoxicillin 500 Mg

INTERVENTIONS:
Drug: Co-Amoxiclav — amoxicillin + clavulanic acid orally
Drug: Paracetamol — paracetamol orally
  Arms: Co-Amoxiclav preoperatively with Metronidazole postoperatively; Co-Amoxiclav preoperatively with amoxicillin postoperatively
Drug: Chlorhexidine mouthwash — 0.2% chlorhexidine mouthwash
Drug: Normal saline — 0.9% normal saline irrigation
Drug: Amoxicillin 500 Mg — Amoxicillin 500 orally
  Arms: Co-Amoxiclav preoperatively with amoxicillin postoperatively
Drug: Metronidazole — metronidazole 500 mg orally
  Arms: Co-Amoxiclav preoperatively with Metronidazole postoperatively

SUMMARY:
There was no evidence to judge the effects of preventative antibiotics for extractions of severely decayed teeth, teeth in diseased gums, or extractions in patients who are sick or have low immunity to infection. Undertaking research in these groups of people may not be possible or ethical. However, it is likely that in situations where patients are at a higher risk of infection that preventative antibiotics may be beneficial, because infections in this group are likely to be more frequent and more difficult to treat To the best of knowledge, no adult study has compared the effects of single dose of Co-Amoxiclave and full oral course before or after dentoalveolar surgery. The current study has formally considered this comparison as a potential valuable trail for reducing the postoperative complications in adult patients who have had surgical removal of teeth under LA.

DETAILED DESCRIPTION:
A comparison of single preoperative dose of Co-amoxiclav versus postoperative full course of Amoxicillin/ Co-amoxiclav in prevention of postoperative complications in dentoalveolar surgery: a randomized controlled trial

Background considerations Prophylactic antibiotics and corticoid in a single dose regimen did not bring any benefit on mandibular third molar surgeries.

Tooth extraction is a surgical treatment to remove teeth that are affected by decay or gum disease or impacted wisdom teeth or those causing pain or inflammation.

The risk of infection after extracting wisdom teeth from healthy young people is about 10%; however, it may be up to 25% in patients who are already sick or have low immunity. Infectious complications include swelling, pain, pus drainage, fever, and also dry socket. Treatment of these infections is generally simple and involves patients receiving antibiotics and drainage of infection from the wound.

A review study was carried out to investigate the effectiveness of Antibiotics to prevent complications following tooth extractions. The findings revealed that there is evidence that prophylactic antibiotics reduce the risk of infection, dry socket and pain following third molar extraction and result in an increase in mild and transient adverse effects. However, patients at a higher risk of infection are more likely to benefit from prophylactic antibiotics, because infections in this group are likely to be more frequent, associated with complications and be more difficult to treat.

Dry socket is a complication that occurs frequently after tooth extraction, causing discomfort to the patient, pain, and a fetid odor. Another study was carried out to investigatethe incidence and risk factors which played the main role in dry socket following surgical removal of impacted third molar in an Iranian population. The outcome of this study revealed that the incidence of dry socket was 19.14%. Age, gender, systemic disorder, and antibiotics use prior to surgery revealed no significant associations with dry socket. However, incidence of dry socket was significantly relevant to smoking, oral contraceptive use, menstruation cycle, difficulty of the surgery according to pre-surgery radiograph evaluation and perception of surgeon post-surgery, length of surgery, and number of carpules used to reach anesthesia. Tolstunov's study demonstrated that the post-extraction socket bleeding is very important for the proper uncomplicated socket healing. If the irrigation solution has not used at the end of extraction, the normal blood clot has a higher likelihood to form, and therefore, can potentially lead to an uncomplicated socket healing without development of alveolar osteitis. Socket bleeding at the extraction site creates a favorable environment for the formation of a blood clot - a protective dressing - necessary for a favorable osseous healing of the socket.

There was no evidence to judge the effects of preventative antibiotics for extractions of severely decayed teeth, teeth in diseased gums, or extractions in patients who are sick or have low immunity to infection. Undertaking research in these groups of people may not be possible or ethical. However, it is likely that in situations where patients are at a higher risk of infection that preventative antibiotics may be beneficial, because infections in this group are likely to be more frequent and more difficult to treat.

To the best of knowledge, no adult study has compared the effects of single dose of Co-Amoxiclave and full oral course before or after dentoalveolar surgery. The current study has formally considered this comparison as a potential valuable trail for reducing the postoperative complications in adult patients who have had surgical removal of teeth under LA.

Primary aim The aim of this study was to assess the efficacy of a single prophylactic dose of Co-Amoxiclave and full oral course in preventing postoperative complications (PC) after a surgical removal of upper and lower teeth.

Material and methods This randomized double-blind clinical trial included 50 patients diagnosed with dentoalveolar surgery. Patients received either preoperative single dose of 625mg Co-Amoxiclav and 1g paracetamol associated with 0.2% chlorhexidine mouthwash or postoperative full course of Co-Amoxiclav for 5 days with 0.9% normal saline irrigation or postoperative full course of amoxicillin 500 mg for five days with 0.9% normal saline irrigation. Patients were reviewed 5 days following the surgery and evaluated if they had alveolar infection, alveolar osteitis, trismus, edema and pain. Difficulty of surgery was reported by the surgeon by using (VAS).

Forty five patients who satisfy the inclusion criteria will be involved in the study and undergo surgical removal of their teeth. . Patients refusing the preoperative dose of oral co-amoxiclav, and unwilling to take part were excluded. Patients who are allergic either to co-amoxiclve or amoxicillin were also excluded. To be included in the study, the tooth must need surgery and require an osteotomy for extraction with use of a motorised drill. Patients will be divided in 3 groups according to the follow up protocol. Patients will be randomly allocated to one of three groups. Patients and assessor will not be aware of the exact treatment which will carry out.

* Treatment 1: 0.9% normal saline irrigation immediately after the surgery with course of Co-Amoxiclav 625 mg 0.2% chlorhexidine mouthwash following the surgery for 5 days (control group)
* Treatment 2: 625 mg Co-Amoxiclav and 1g Paracetamol preoperatively and 0.2% chlorhexidine mouthwash immediately before the surgery with course of Metronidazole 500 mg and 0.2% chlorhexidine mouthwash following the surgery for 5 days
* Treatment 3: 625 mg Co-Amoxiclav and 1g Paracetamol preoperatively and 0.2% chlorhexidine mouthwash immediately before the surgery with course of amoxicillin 500 mg and 0.2% chlorhexidine mouthwash following the surgery for 5 days

All surgeries will be done under local anaesthesia. A standard extraction technique of surgery will be employed for the patient in first group. This include a buccal full-thickness flap, buccal trough (osteotomy) and extraction of the tooth), followed by a traditional end-of-surgery debridement protocol consisting of a gentle curettage, socket irrigation with approximately 5 ml of sterile normal saline solution , socket suctioning and placement of stitches.

* Signs of alveolar osteitis may include:

  1. An empty socket, which is partially or totally devoid of blood clot.
  2. Exposed bone may be visible or the clot may be filled with food debris which reveals the exposed bone once it is removed. The exposed bone is extremely painful to touch.
  3. Surrounding inflamed soft tissues may overlie the socket and hide the dry socket from casual examination (Daly et al., 2012)
* Symptomsof alveolar osteitis may include:

  1. Dull, aching, throbbing pain in the area of the socket, which is moderate to severe and may radiate to other parts of the head such as the ear, temple and neck. The pain normally starts on the second to fourth day after the extraction,[ and may last 10-40 days.The pain may be so strong that even strong analgesics do not relieve it.
  2. Intraoral halitosis
  3. Bad taste in the mouth (Fragiskos, 2007)
* Signs and symptoms of oral infection

  1. Oral swelling
  2. Tenderness with touch
  3. Pus drainage
  4. Difficulty fully opening your mouth or swallowing. Power calculation A study with 45 subjects was reported to have 90% power to detect a difference in success rate of 21% (Bortoluzzi et al, 2013) in a continuous outcome measure assuming a significance level of 5% and a correlation of 0.5 between responses from the different subjects.

ELIGIBILITY:
Inclusion Criteria:

* Patient age from 16 to 70 yrs old
* Patient needs surgical teeth extraction (subject tooth will be removed using osteotomy by motorised drill).

Exclusion Criteria:

* Patients refusing the preoperative dose of oral co-amoxiclav, and unwilling to take part .
* Patients who are allergic to co-amoxiclve, amoxicillin or metronidazole
* Patient are on warfarin medication

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2019-10-02 (Actual); Primary Completion 2020-12-02 (Estimated); Study Completion 2021-01-20 (Estimated)

PRIMARY OUTCOMES:
infection rate | 5 days after extraction assessment
  dry socket after surgical extraction

CONTACTS AND LOCATIONS:
Locations (1):
- Taibah University, Madinah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes